CLINICAL TRIAL: NCT03367702
Title: Phase III IGRT and SBRT vs IGRT and Hypofractionated IMRT for Localized Intermediate Risk Prostate Cancer
Brief Title: Stereotactic Body Radiation Therapy or Intensity-Modulated Radiation Therapy in Treating Patients With Stage IIA-B Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: NRG Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRG-GU005; NCI-2017-01398 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GU005 (Other: NRG Oncology); NRG-GU005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Stage II Prostate Adenocarcinoma AJCC v7
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (IMRT) (Active Comparator): Patients undergo IMRT once daily for 5 fractions per week for 20 or 28 fractions over less than 32 business days.
  Interventions: Radiation: Intensity-Modulated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (SBRT) (Experimental): Patients undergo SBRT at least every other day for 2-3 fractions per week over less than 17 business days.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
  Arms: Arm I (IMRT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Arm II (SBRT)

SUMMARY:
This randomized phase III trial studies how well stereotactic body radiation therapy works compared to intensity-modulated radiation therapy in treating patients with stage IIA-B prostate cancer. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Stereotactic body radiation therapy may work better in treating patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether stereotactic body radiation therapy (SBRT) can be shown to be superior to hypofractionated intensity-modulated radiation therapy (IMRT) in terms of genitourinary (GU) and gastrointestinal (GI) toxicity by having fewer patients that experience a minimal important decline (MID) in urinary irritation/obstructive and bowel Health Related Quality of Life (HRQOL) as measured by Expanded Prostate Cancer Index Composite (EPIC)-26 at 24 months post completion of therapy.

II. To determine if SBRT (5 fractions of 7.25 Gy) is superior to hypofractionated IMRT (28 fractions of 2.5 Gy or 20 fractions of 3 Gy) as measured by disease free survival (DFS).

SECONDARY OBJECTIVES:

I. To determine whether SBRT can be shown to be superior to hypofractionated IMRT at 12 and 24 months post completion of therapy in terms of HRQOL by having fewer patients that experience a minimal important decline (MID) bowel (12 months only) sexual, hormonal, urinary irritation/obstructive (12 months only) and in urinary incontinence HRQOL as measured by EPIC-26.

II. To determine if SBRT (5 fractions of 7.25 Gy) is superior to hypofractionated IMRT (28 fractions of 2.5 Gy or 20 fractions of 3 Gy) as measured by biochemical failure, overall survival, local failure, prostate cancer specific survival, and distant metastases.

III. To determine the correspondence between the diagnostic magnetic resonance imaging (MRI) and biopsy.

IV. To determine if prostate imaging-reporting and data system (PIRADS)version (v)2.1 = 4/5 disease is prognostic for biochemical failure.

EXPLORATORY OBJECTIVES:

I. To determine whether a potentially more expensive therapy, SBRT, would be cost-effective than standard hypofractionated IMRT as measured by the European Quality of Life Five Dimension Five Level Scale Questionnaire (EQ-5D-5L).

II. To determine if disease characteristics captured on baseline and follow-up MRI can be used to predict which patients will respond to SBRT versus hypofractionated IMRT.

III. To validate autosegmentation tools for the prostate and tumors. IV. Collect specimens for future translational research analyses.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients undergo IMRT once daily for 5 fractions per week for 20 or 28 fractions over less than 32 business days.

ARM II: Patients undergo SBRT at least every other day for 2-3 fractions per week over less than 17 business days.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated (no local therapy such as surgery, radiation cryotherapy, high-intensity focused ultrasound [HIFU], etc.) localized adenocarcinoma of the prostate with the following clinical findings:

  * Clinical stage by digital rectal exam of either T1c or T2a/b (limited to one side of the gland); (American Joint Committee on Cancer [AJCC], version 7) or cT1a-c or 2a or 2b
  * Stages T1a-T1b are eligible if patient underwent transurethral prostatic resection (TURP)
  * The patient must meet one of the following 3 criteria: 1) Gleason score must be Gleason 7(3+4) with a PSA < 20 ng/mL, or 2) Gleason 6 (3+3) with a PSA > 10 ng/mL and < 20 ng/mL which is considered intermediate risk and eligible for the study (AJCC, version 7), or 3) Group Grade 1 with a PSA > 10 ng/mL and < 20 ng/mL or 2 with a PSA < 20 ng/mL

    * If patient is receiving a 5-alpha reductase inhibitor at the time of enrollment, the baseline PSA value may be double the initial value and the medication should be discontinued but a washout period is not required; to be eligible, a PSA drawn while still on the medicine must be:

      * < 10 ng/mL if Gleason 7(3+4) (note this patient would be on stratification level 1 if PSA < 5 ng/mL and stratification level 2 if less than 10 ng/mL)
      * > 5 ng/mL and less than 10 ng/mL for Gleason 6(3+3) (note this patient would be on stratification level 3)
  * The prostate volume must be < 70 cc as reported at time of biopsy or by separate measure with ultrasound or other imaging modalities including magnetic resonance imaging (MRI) or computed tomography (CT) scan
  * Patients in active surveillance who elect to be treated are eligible if they meet protocol requirements
* Age >= 18
* History and physical including a digital rectal exam 60 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 60 days prior to registration
* MRI of the prostate and pelvis (per institutional standard of care [SOC] - should be compliant with PIRADSv2.1 guidelines) within 1 year prior to registration
* Bone scan as clinically indicated within 120 days prior to registration
* Charlson modified co-morbidity score =< 4 for patients under 60 and =< 5 for patients 60 and over 21 days prior to registration
* International prostate symptom score (IPSS) of < 15 21 days prior to registration
* The patient must provide study-specific informed consent prior to study entry
* Willingness and ability to complete the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaire
* Completion of all items of the EPIC-26 which will be data entered at registration 60 days prior to registration
* Only English, Spanish, and French-speaking patients are eligible to participate as these are the only languages EPIC-26 has been validated in

Exclusion Criteria:

* Definitive clinical or radiologic evidence of metastatic disease; no nodal involvement or evidence of metastatic disease allowed as defined by screening of the pelvis
* Definitive T3 disease on MRI
* Prior or current invasive malignancy with current evidence of active disease within the past 2 years

  * Exceptions: Non-melanomatous skin cancer, carcinoma in situ of the male breast, penis, oral cavity, or stage Ta of the bladder, or stage I completely resected melanoma
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable; must be off treatment for at least 3 years
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* The use of hormonal therapy is not allowed; if the patient is on a 5-alpha reductase inhibitor, then they should be stopped prior to treatment once enrolled onto the study; no washout period is required for this study to participate
* Severe, active co-morbidity defined as follows:

  * Human immunodeficiency virus (HIV) positive with CD4 count < 200 cells/microliter; Note that patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count >= 200 cells/microliter within 30 days prior to registration; Note also that HIV testing is not required for eligibility for this protocol; this exclusion criterion is necessary because the treatments involved in this protocol may be significantly immunosuppressive
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol; (patients on Coumadin or other blood thinning agents are eligible for this study)
* Contraindication to MRI

  * Cardiac pacemaker or defibrillator
  * Surgically implanted electrical devices such as spinal stimulation devices or intracranial stimulation devices, cochlear implants, the presence of metallic foreign bodies in the orbits, and incompatible old mechanical heart valves and aneurysm clips

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients-reported gastrointestinal and genitourinary toxicity | Up to 2 years
  Will be measured by Expanded Prostate Cancer Index Composite-(EPIC) 26 bowel and urinary irritation domains. Will be compared between treatment arms using a test of proportions with two-sided significance level of 0.05.
Disease free survival | Time to biochemical failure (Phoenix definition), local failure, regional failure, distant metastasis, or death from any cause, assessed up to 2 years
  Will be estimated using the Kaplan-Meier method and treatment arms compared using the stratified log-rank test.

SECONDARY OUTCOMES:
Health related quality of life | Up to 2 years
  Will be measured by EPIC-26 urinary incontinence, sexual, and hormonal domains.
Biochemical failure | Up to 2 years
  Will be assessed by Phoenix definition.
Local failure | From the time of randomization to the date of local failure, date of precluding death, or last known follow-up date, assessed for up to 2 years
Regional failure | From the time of randomization to the date of local failure, date of precluding death, or last known follow-up date, assessed for up to 2 years
Distant metastasis | From the time of randomization to the date of distant metastasis, date of precluding death, or last known follow-up date, assessed for up to 2 years
Prostate cancer specific survival | Up to 2 years
Overall survival | From the date of randomization to the date of death or last known follow-up date, with patients alive at the last known follow-up time treated as censored, assessed up to 5 years
  Will be estimated using the Kaplan-Meier method and treatment arms compared using the stratified log-rank test.
Incidence of adverse events (AEs) | Up to 2 years
  Will be assessed by Common Terminology Criteria for Adverse Events version 5.0. Counts of all AEs by grade will be provided by treatment arm. Counts and frequencies will be provided for the worst grade AE experienced by the patient by treatment arm. The number of patients with at least 1 grade 3 or higher AE will be compared between the treatment arms. A comparison between treatment arms of grade 3 and higher genitourinary (GU) and gastrointestinal (GI) events related to treatment (separately) will also be tested. There are 5 pre-specified AEs, dysuria, hematuria, incontinence, rectal bleeding, and fatigue. A comparison of any event and grade and higher events will be compared between treatment arms. All comparisons will be tested using a Chi-Square test with a significance level of 0.05.
Presence of Prostate Imaging-Reporting and Data System version (PIRADSv) 2 = 4/5 disease | Baseline
  Will be assessed by magnetic resonance imaging (MRI).
Predictive value of PIRADSv2 = 4/5 disease for biochemical failure | Up to 2 years
  Predictive value of PIRADSv2 = 4/5 disease for biochemical failure

OTHER OUTCOMES:
Central manual user segmentation of tumors | Up to 2 years
  Central manual user segmentation of tumors
Performance of supervised automated tumor detection toolset | Up to 2 years
  Performance of supervised automated tumor detection toolset
Performance of supervised automated tumor segmentation toolset | Up to 5 years
  Performance of supervised automated tumor segmentation toolset
Image registration performance | Up to 2 years
  Image registration performance
Predictive utility of radiomic analysis | Up to 2 years
  Predictive utility of radiomic analysis
Predictive value for local control and biochemical failure | At 2 years
  Will be assessed by MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Rodney J Ellis, Principal Investigator — NRG Oncology
Locations (293):
- United States (276):
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - Lewis and Faye Manderson Cancer Center, Tuscaloosa, Alabama
  - Arizona Center for Cancer Care - Gilbert, Gilbert, Arizona
  - Arizona Center for Cancer Care-Peoria, Peoria, Arizona
  - Arizona Center for Cancer Care - Scottsdale, Scottsdale, Arizona
  - Arizona Center for Cancer Care-Surprise, Surprise, Arizona
  - Arizona Oncology Associates-West Orange Grove, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Fresno Cancer Center, Fresno, California
  - Marin General Hospital, Greenbrae, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Woodland Memorial Hospital, Woodland, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - GenesisCare USA - Key West, Key West, Florida
  - GenesisCare USA - Lakewood Ranch, Lakewood Rch, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - GenesisCare USA - Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Edward Hines Jr VA Hospital, Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Midwestern Regional Medical Center, Zion, Illinois
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Parkview Regional Medical Center, Fort Wayne, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Central Maryland Radiation Oncology in Howard County, Columbia, Maryland
  - University of Maryland Shore Medical Center at Easton, Easton, Maryland
  - UM Baltimore Washington Medical Center/Tate Cancer Center, Glen Burnie, Maryland
  - TidalHealth Richard A Henson Cancer Institute, Ocean Pines, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Mass General/North Shore Cancer Center, Danvers, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Michigan Healthcare Professionals Clarkston, Clarkston, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Michigan Healthcare Professionals Farmington, Farmington Hills, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Michigan Healthcare Professionals Macomb, Macomb, Michigan
  - Michigan Healthcare Professionals Madison Heights, Madison Heights, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Michigan Healthcare Professionals Troy, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - SSM Health Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Exeter Hospital, Exeter, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Saint Peter's Health Partners, Albany, New York
  - New York-Presbyterian/Brooklyn Methodist Hospital, Brooklyn, New York
  - Sands Cancer Center, Canandaigua, New York
  - Mary Imogene Bassett Hospital, Cooperstown, New York
  - Garnet Health Medical Center, Middletown, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Scotland Memorial Hospital-Laurinburg Cancer Center, Laurinburg, North Carolina
  - Duke Cancer Center Raleigh, Raleigh, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Geauga Hospital, Chardon, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - The Radiation Oncology Center-Hilton Head/Bluffton, Hilton Head Island, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Texas Cancer Center, Abilene, Texas
  - Texas Oncology-McKinney, McKinney, Texas
  - Texas Oncology-Plano West, Plano, Texas
  - Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Deke Slayton Cancer Center, Webster, Texas
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Sentara Cancer Institute at Sentara CarePlex Hospital, Hampton, Virginia
  - Bon Secours DePaul Medical Center, Norfolk, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Roanoke, Virginia
  - Sentara Obici Hospital, Suffolk, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
- Canada (12):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Centre De Sante Et De Services Sociaux De Chicoutimi, Chicoutimi, Quebec
  - CIUSSSEMTL-Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Research Institute of the McGill University Health Centre (MUHC), Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke-Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Chai Wan, Hong Kong
- Tata Memorial Hospital, Mumbai, India
- Ireland (2):
  - Beacon Hospital, Dublin, Co Dublin
  - Saint Lukes Hospital, Dublin, Co Dublin
- Kantonsspital Aarau, Aarau, Switzerland

REFERENCES:
- [Derived] Alley S, Tonneau M, Olivie D, Tempany-Afdhal CM, Choyke PL, Turkbey IB, van der Heide UA, Ellis RJ, Kadoury S, Boike TP, Pennington JD, Frazier A, Lawton CAF, Leong N, Mihai AM, Morgan SC, Solanki AA, Michalski JM, Feng FY, Sandler HM, Menard C. Assessing Quality and Adherence to PI-RADSv2.1 Minimum Technical Standards of Prostate MRI in NRG-GU005. J Magn Reson Imaging. 2026 Feb;63(2):464-474. doi: 10.1002/jmri.70142. Epub 2025 Oct 8. PMID 41063518
- [Derived] Alley S, Jackson E, Olivie D, Van der Heide UA, Menard C, Kadoury S. Effect of magnetic resonance imaging pre-processing on the performance of model-based prostate tumor probability mapping. Phys Med Biol. 2022 Dec 13;67(24). doi: 10.1088/1361-6560/ac99b4. PMID 36223780